CLINICAL TRIAL: NCT02189759
Title: A Randomized Trial of Kangaroo Mother Care to Prent Neonatal Hypothermia - Trials 2A & 2 B
Brief Title: Kangaroo Mother Care to Prevent Hypothermia in Term Infants
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Responsible Party: Principal Investigator, Manimaran Ramani, MD, Assistant Professor of Pediatrics, University of Alabama at Birmingham
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: UAB Neo 012
Record Dates: First submitted 2014-07-11; First posted 2014-07-15 (Estimated); Results first posted 2017-06-19 (Actual); Last update posted 2017-06-19 (Actual); Status verified 2017-04

CONDITIONS: Hypothermia; Newborn
Keywords: Hypothermia; Hyperthermia; Kangaroo Mother Care; Newborn
MeSH Terms: conditions — Hypothermia; Hyperthermia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Continuous Kangaroo Mother Care to one hour after birth (Active Comparator): In addition to standard WHO thermoregulation care which includes warm delivery rooms, immediate drying, Kangaroo Mother Care (KMC) whenever possible, early and exclusive breastfeeding, postponed bathing and weighing if needed, appropriate bundling and placing the infant in air incubator, radiant heater, or heat mattress if the infant develops hypothermia, the infants will receive continuous KMC most of the time possible from birth to one hour after birth.
  Interventions: Other: Continuous Kangaroo Mother Care to one hour after birth
- Standard Kangaroo Mother Care to one hour after birth (Sham Comparator): Infants will receive standard WHO thermoregulation care which includes warm delivery rooms, immediate drying, Kangaroo Mother Care (KMC) whenever possible, early and exclusive breastfeeding, postponed bathing and weighing if needed, appropriate bundling and placing the infant in air incubator, radiant heater, or heat mattress if the infant develops hypothermia from birth to 1 hour after birth.
  Interventions: Other: Standard Kangaroo Mother Care to one hour after birth
- Continuous Kangaroo Mother Care to discharge (Active Comparator): In addition to standard WHO thermoregulation care which includes warm delivery rooms, immediate drying, Kangaroo Mother Care (KMC) whenever possible, early and exclusive breastfeeding, postponed bathing and weighing if needed, appropriate bundling and placing the infant in air incubator, radiant heater, or heat mattress if the infant develops hypothermia, the infants will receive continuous KMC most of the time possible from one hour after birth to discharge.
  Interventions: Other: Continuous Kangaroo Mother Care to discharge
- Standard Kangaroo Mother Care to discharge (Sham Comparator): Infants will receive standard WHO thermoregulation care which includes warm delivery rooms, immediate drying, Kangaroo Mother Care (KMC) whenever possible, early and exclusive breastfeeding, postponed bathing and weighing if needed, appropriate bundling and placing the infant in air incubator, radiant heater, or heat mattress if the infant develops hypothermia from 1 hour after birth to discharge.
  Interventions: Other: Standard Kangaroo Mother Care to discharge

INTERVENTIONS:
Other: Continuous Kangaroo Mother Care to one hour after birth — Infants will receive the standard WHO thermoregulation care with encouragement from study personnel to keep infant in Kangaroo Mother Care for as much as possible until 1 hour of birth. In KMC, the naked newborn infant with cap and diaper will be placed prone on mom's bare chest with blanket covering infant's back. All infants will be resuscitated as usual per Neonatal Resuscitation Program guidelines and hospital standard practices. The nursing staff will supervise mother-infant when mother is sleeping with infant in KMC. If infant becomes hyperthermic (>38 degrees Celsius), the infant will be removed from KMC and routine bundling practices will be used. The infant's temperature will be taken via axillae with a digital thermometer at one hour of age.
  Arms: Continuous Kangaroo Mother Care to one hour after birth
Other: Standard Kangaroo Mother Care to one hour after birth — Infants will receive the standard WHO thermoregulation care of Kangaroo Mother Care for as much as possible until 1 hour of birth, without additional encouragement per study personnel. In KMC, the naked newborn infant with cap and diaper will be placed prone on mom's bare chest with blanket covering the infant's back. All infants will be resuscitated as usual per Neonatal Resuscitation Program guidelines and hospital standard practices. The nursing staff will supervise mother-infant when mother is sleeping with infant in KMC. If infant becomes hyperthermic (>38 degrees Celsius), the infant will receive standard care which may include removal from KMC and use of routine bundling practices. The infant's temperature will be taken via axillae with a digital thermometer at one hour of age.
  Arms: Standard Kangaroo Mother Care to one hour after birth
Other: Continuous Kangaroo Mother Care to discharge — Infants will receive the standard WHO thermoregulation care with encouragement from study personnel to keep infant in Kangaroo Mother Care for as much as possible from one hour after birth to discharge. In KMC, the naked newborn infant with cap and diaper will be placed prone on mom's bare chest with blanket covering the infant's back. The nursing staff will supervise mother-infant when mother is sleeping with infant in KMC. If infant becomes hyperthermic (>38 degrees Celsius), the infant will be removed from KMC and routine bundling practices will be used. The infant's temperature will be taken via axillae with a digital thermometer at one hour of age and again at discharge or 24 hours whichever occurs first.
  Arms: Continuous Kangaroo Mother Care to discharge
Other: Standard Kangaroo Mother Care to discharge — Infants will receive the standard WHO thermoregulation care without additional encouragement from study personnel to keep infant in Kangaroo Mother Care for as much as possible from 1 hour after birth to discharge. In KMC, the naked newborn infant with cap and diaper will be placed prone on mom's bare chest with blanket covering the infant's back. The nursing staff will supervise mother-infant when mother is sleeping with infant in KMC. If infant becomes hyperthermic (>38 degrees Celsius), standard treatment will be given which may include removal from KMC and use of routine bundling practices. The infant's temperature will be taken via axillae with a digital thermometer at one hour of age and again at discharge or 24 hours whichever occurs first.
  Arms: Standard Kangaroo Mother Care to discharge

SUMMARY:
The overall hypothesis is that better adherence to Kangaroo Mother Care (KMC) in combination with existing WHO thermoregulation care will reduce the incidence of moderate hypothermia (32-36 degrees C) or severe hypothermia (<32.0 degrees C) in term infants (greater than or equal to 37 weeks of gestational age) when compared with routine WHO thermoregulation alone.

DETAILED DESCRIPTION:
The overall hypothesis is that better adherence to Kangaroo Mother Care (KMC) in combination with existing World Health Organization (WHO) thermoregulation care (warm delivery rooms, immediate drying after birth, KMC whenever possible, early and exclusive breastfeeding, postponement of bathing and weighing, appropriate bundling, and use of air incubator, radiant warmer, or heat mattress if the neonate develops hypothermia) will reduce the incidence of moderate hypothermia (32-36 degrees C) or severe hypothermia (<32.0 degrees C) in term infants (greater than or equal to weeks of gestational age) when compared with routine WHO thermoregulation alone.

ELIGIBILITY:
Inclusion Criteria:

* Estimated gestational age greater than or equal to 37 weeks
* Delivery in the hospital

Exclusion Criteria:

* Abdominal wall defect or myelomeningocele
* Major congenital anomalies
* Blistering skin disorder

Ages: 1 Minute to 2 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 375 (Actual)
Dates: Start 2014-08 (Actual); Primary Completion 2014-09 (Actual); Study Completion 2014-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Waldemar A Carlo, MD, Study Director — University of Alabama at Birmingham; Manimaran Ramani, MD, Principal Investigator — University of Alabama at Birmingham
Locations (1):
- University Teaching Hospital, Lusaka, Zambia

REFERENCES:
- [Derived] Ramani M, Choe EA, Major M, Newton R, Mwenechanya M, Travers CP, Chomba E, Ambalavanan N, Carlo WA. Kangaroo mother care for the prevention of neonatal hypothermia: a randomised controlled trial in term neonates. Arch Dis Child. 2018 May;103(5):492-497. doi: 10.1136/archdischild-2017-313744. Epub 2018 Feb 22. PMID 29472198

RESULTS

PARTICIPANT FLOW:
Groups:
- Continuous Kangaroo Mother Care to One Hour After Birth: Continuous Kangaroo Mother Care to one hour after birth: Infants will receive the standard WHO thermoregulation care with encouragement from study personnel to keep infant in Kangaroo Mother Care for as much as possible until 1 hour of birth. In KMC, the naked newborn infant with cap and diaper will be placed prone on mom's bare chest with blanket covering infant's back. All infants will be resuscitated as usual per Neonatal Resuscitation Program guidelines and hospital standard practices. The nursing staff will supervise mother-in
- Standard Kangaroo Mother Care to One Hour After Birth: Standard Kangaroo Mother Care to one hour after birth: Infants will receive the standard WHO thermoregulation care of Kangaroo Mother Care for as much as possible until 1 hour of birth, without additional encouragement per study personnel. In KMC, the naked newborn infant with cap and diaper will be placed prone on mom's bare chest with blanket covering the infant's back. All infants will be resuscitated as usual per Neonatal Resuscitation Program guidelines and hospital standard practices. The nursing staff will supervise mother-infant when mother is sleeping with infant in KMC. If infant bec
- Continuous Kangaroo Mother Care to Discharge: Continuous Kangaroo Mother Care to discharge: Infants will receive the standard WHO thermoregulation care with encouragement from study personnel to keep infant in Kangaroo Mother Care for as much as possible from one hour after birth to discharge. In KMC, the naked newborn infant with cap and diaper will be placed prone on mom's bare chest with blanket covering the infant's back. The nursing staff will supervise mother-infant when mother is sleeping with infant in KMC. If infant becomes hyperthermic (>38 degrees Celsius), the
- Standard Kangaroo Mother Care to Discharge: Standard Kangaroo Mother Care to discharge: Infants will receive the standard WHO thermoregulation care without additional encouragement from study personnel to keep infant in Kangaroo Mother Care for as much as possible from 1 hour after birth to discharge. In KMC, the naked newborn infant with cap and diaper will be placed prone on mom's bare chest with blanket covering the infant's back. The nursing staff will supervise mother-infant when mother is sleeping with infant in KMC. If infant becomes hyperthermic (>38 degrees Celsius), standard treatment will be given which may include remova
Period: Overall Study
Arm/Group | Continuous Kangaroo Mother Care to One Hour After Birth | Standard Kangaroo Mother Care to One Hour After Birth | Continuous Kangaroo Mother Care to Discharge | Standard Kangaroo Mother Care to Discharge
Started | 102 | 101 | 83 | 89
Completed | 102 | 101 | 81 | 84
Not Completed | 0 | 0 | 2 | 5
Not completed — Lost to Follow-up | 0 | 0 | 2 | 5

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Continuous Kangaroo Mother Care to One Hour After Birth | Standard Kangaroo Mother Care to One Hour After Birth | Continuous Kangaroo Mother Care to Discharge | Standard Kangaroo Mother Care to Discharge | Total
Number analyzed (Participants) | 102 | 101 | 81 | 84 | 368
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 102 | 101 | 81 | 84 | 368
  Between 18 and 65 years | 0 | 0 | 0 | 0 | 0
  >=65 years | 0 | 0 | 0 | 0 | 0
Age, Continuous [Mean (Full Range); unit: hours] | 1 [.5 to 1] | 1 [.5 to 1] | 6 [1 to 12] | 6 [1 to 12] | 6 [1 to 12]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 52 | 54 | 42 | 46 | 194
  Male | 50 | 47 | 39 | 38 | 174
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 102 | 101 | 81 | 84 | 368
  White | 0 | 0 | 0 | 0 | 0
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  Zambia | 102 | 101 | 81 | 84 | 368

OUTCOME MEASURES:

1. Primary Outcome: Number of Infants With Axillary Temperature <36.0 Degrees Celsius
Description: Temperature taken per axilla using digital thermometer
Time Frame: Time of birth to 1 hour
Measure: Count of Participants; unit: Participants
Arm/Group | Continuous Kangaroo Mother Care to One Hour After Birth | Standard Kangaroo Mother Care to One Hour After Birth
Number analyzed (Participants) | 102 | 101
Participants | 55 | 56

2. Primary Outcome: Number of Infants With Axillary Temperature < 36.0 Degrees Celsius at Discharge
Description: Temperature taken per axilla using diigital thermometer at Discharge or 24hrs after birth
Time Frame: At discharge or 24 hours after birth (whichever is first)
Measure: Count of Participants; unit: Participants
Arm/Group | Continuous Kangaroo Mother Care to Discharge | Standard Kangaroo Mother Care to Discharge
Number analyzed (Participants) | 81 | 84
Participants | 14 | 14

3. Secondary Outcome: Number Infants Admitted to the Neonatal Intensive Care Unit
Description: Any admission to the neonatal intensive care unit for higher level care
Time Frame: Duration of hospitalization-an average of 2 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Continuous Kangaroo Mother Care to One Hour After Birth | Standard Kangaroo Mother Care to One Hour After Birth | Continuous Kangaroo Mother Care to Discharge | Standard Kangaroo Mother Care to Discharge
Number analyzed (Participants) | 102 | 101 | 81 | 84
Participants | 0 | 0 | 0 | 0

4. Secondary Outcome: Duration of Kangaroo Mother Care
Description: Skin to skin contact between baby and mother
Time Frame: Duration of hospitalization-an average of 2 weeks
Population: Infants in "Standard Kanagroo Mother Care to one hour after birth" and "Standard Kangaroo Mother care to discharge" groups received kangaroo mother care only during breastfeeding
Measure: Mean (Standard Error); unit: Hours
Arm/Group | Continuous Kangaroo Mother Care to One Hour After Birth | Standard Kangaroo Mother Care to One Hour After Birth | Continuous Kangaroo Mother Care to Discharge | Standard Kangaroo Mother Care to Discharge
Number analyzed (Participants) | 102 | 101 | 81 | 84
Hours | .6 (.25) | 0 (0) | 7 (4) | 0 (0)

ADVERSE EVENTS:
Description: All-Cause Mortality, Serious, and Other [Not Including Serious] Adverse Events were not monitored/assessed
Arm/Group | Continuous Kangaroo Mother Care to One Hour After Birth | Standard Kangaroo Mother Care to One Hour After Birth | Continuous Kangaroo Mother Care to Discharge | Standard Kangaroo Mother Care to Discharge
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0 | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No